CLINICAL TRIAL: NCT04863352
Title: Health Status, Quality of Life and Function in Survivors After Radical Treatment for Prostate Cancer. A Cross-sectional Study Focusing on Older Survivors. Part I and IIA
Brief Title: Health Status, Quality of Life and Function in Survivors After Radical Treatment for Prostate Cancer. Part I and IIA
Acronym: OPS
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 150410
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer, radical treatment, radiotherapy, surgery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Men who have been treated for localized or locally advanced prostate cancer with curative intent
- Matched population based controls: Existing population based data from men who participated in the Trøndelag Health Survey 2017-2019

SUMMARY:
In this study, addressing prostate cancer survivors, i.e. men who received potentially curative (radical) treatment two to six years ago, we will investigate if older age at time of treatment is a detrimental factor with respect to long-term quality of life (Qol), health, and function. We will also compare QoL, health and function between the prostate cancer survivors and matched population based cohorts, and thereby provide realistic information on the long-term impact of radical prostate cancer treatment

DETAILED DESCRIPTION:
Prostate cancer is the most common male cancer in Norway, with almost 5000 new cases yearly. More than12 % of men contract prostate cancer before the age of 75. As 5-year survival is high (>95%), a significant proportion of the older male population are prostate cancer survivors. The quality of life (QoL) and daily function of these older males need elucidation to provide adequate health care services and information to this large patient group.

The present project includes two studies(Study I and IIA). Study I is investigating the QoL, health status, and local adverse treatment effects in all men 2-6 years after radical treatment for prostate cancer. Local adverse treatment effects are defined as problems related to organs and structures adjacent to the prostate gland (e.g. bowel and urinary problems, and sexual dysfunction). Study IIA will focus on older prostate cancer survivors, defined as men who were 70 years or older by the time of treatment. To complete the overall project, we also plan a later study, Study IIB, that will investigate in more detail the physical functioning and performance of the older survivors.

Design Study I: A cross-sectional survey targeting all patients from the catchment area of Innlandet Hospital Trust (SI-HF) who received radical treatment for localized/locally advanced prostate cancer at SI-HF from 2014 to 2018 Study II A: A supplementary cross-sectional survey targeting older participants from Study I who were >70 years at time of treatment Control groups: For comparison with a general population, we will use existing data from male participants in the fourth wave of the Trøndelag Health Study (HUNT4) including the HUNT4 70+ survey. Control groups will be drawn, matched on age and education. HUNT4 and HUNT4 70+ were both performed in 2017-2019, and targeted all inhabitants and inhabitants >70 years respectively in the former Nord-Trøndelag County. Jointly they include broad health assessments using questionnaires, physical examinations, and tests.

Study aims Primary study aims are

1. to investigate if older age at the time of radical treatment has a negative impact on self-reported QoL, function and local adverse effects in prostate cancer survivors
2. to investigate if health status, health problems, and use of health care services in older prostate cancer survivors differ from a general male population of the same age

Secondary aims are

1. to investigate how local adverse effects after radical prostate cancer treatment may influence QoL and functioning in both older and younger survivors, and to explore how other factors such as treatment modality and comorbidity may influence these outcomes
2. to investigate if health status, health problems, and use of health care services in younger prostate cancer survivors (being < 70 years by the time of treatment) differ from a general male population of the same age

Study conduct

All men who are eligible according to the inclusion criteria (see sample size below and inclusion criteria), will be invited to participate. All participants will provide written informed consent.

In Study I, participants will be asked to fill in a questionnaire covering QoL (EORTC QLQ-C30 questionnaire), local adverse effects after prostate cancer treatment (the EPIC-26) and other health problems (selected items from the HUNT4 Survey). Participants in Study I, who were 70 years or more by the time they received their cancer treatment, will subsequently be asked to fill in an additional questionnaire covering a broader range of health issues also with items from the HUNT4 Survey (Study IIA). Questionnaires will be administered by post with pre-paid return envelopes attached.

To fulfill our aims, we will investigate the association between age at treatment and QoL, self-reported health status, and local adverse effects (Primary aim 1). Furthermore, we will compare self-reported health, health problems, and use of health care services between our study population and the drawn control group (Primary aim 2 and Secondary aim 2). We will also investigate how local adverse effects may influence prostate cancer survivors' QoL and functioning (Secondary aim 1).

Sample size and statistics

About 1400 men with prostate cancer received curative treatment for local or localized prostate cancer at Innlandet Hospital Trust from 2014 to 2018, and about 1200 of these are estimated to be eligible for the initial study I. Matched controls will be drawn from the HUNT4 and HUNT4 70+ surveys, distribution 1:3 (cancer survivors : controls).

Simple descriptive statistics will be used to describe our cohorts. Comparison between groups will be made using parametric and non-parametric statistics as appropriate. To assess the impact of age, treatment regimen and relevant confounding factors on outcomes, multiple regression models will be estimated.

ELIGIBILITY:
Inclusion Criteria. Study group:

Study I:

a) men who received radical radiotherapy or robot-assisted radical prostatectomy for prostate cancer at Innlandet Hospital Trust 01.01.2014 and 31.12.2018; b) alive and living in Innlandet County; c) fluent in Norwegian (orally and in writing); provide written informed consent

Study IIa) the subgroup of participants in Study I who were > 70 years by the time of treatment.

Exclusion Criteria: None

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study group: Men who have received radical treatment for prostate cancer at Innlandet Hospital Trust 2014 to 2018
Study Population: Study group: Men having received radical treatment for prostate cancer at Innlandet Hospital Trust, see eligibility criteria
  Control group: For comparison with a general population, a control group of males matched on age and education will be drawn from the Trøndelag Health Survey 4 (HUNT4) and HUNT4 70+ surveys performed in 2017-2019, targeting all inhabitants and inhabitants >70 years in Trøndelag County, respectively
Sampling Method: Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Global quality of life | at time of assessment (cross-sectional)
  Global quality of life assessed by the EORTC QLQ-C30 questionnaire's global QoL scale ranging from 0 to 100, higher scores indicate better QoL
General health | at time of assessment (cross-sectional)
  self-reported using items from the Trøndelag Health Survey 4, categorical scale: bad/not so go good/good/very good

SECONDARY OUTCOMES:
physical function | at assessment (cross-sectional)
  as measured by the EORTC QLQ-C30 questionnaire's physical functioning scale, ranging from 0-100, higher scores indicate better function
EPIC-26 scores | at assessment (cross-sectional)
  Local late effects of prostate cancer treatment as measured by the EPIC-26
Activities of daily living | at assessment (cross-sectional)
  as measured by items from The Trøndelag Health Survey 4

CONTACTS AND LOCATIONS:
Overall Officials: Marit Slaaen, PhD, Study Chair — Sykehuset Innlandet HF; Ola Berger Christiansen, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Brumunddal, Norway

IPD SHARING:
Plan to Share IPD: No
According to Norwegian Privacy Protection regulations, data cannot be shared as long as they are not anonymised. However, insight into all data is possible by visiting our research site

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT04863352/Prot_SAP_000.pdf